CLINICAL TRIAL: NCT05070117
Title: The Effect of Exercise Training on Musculoskeletal Health in Individuals With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Jose State University (Other)
Responsible Party: Principal Investigator, Areum Jensen, Assistant Professor, San Jose State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F17081
Record Dates: First submitted 2021-08-23; First posted 2021-10-07 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance/strength training (Experimental)
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Study participants perform resistance/strength exercises 2-3 times per week for one hour, for one year.

SUMMARY:
Cerebral palsy (CP) is a neurodevelopmental disorder and is the most common childhood disability. CP is characterized by abnormal development, impaired motor function, and muscular and skeletal abnormalities. Due to their diminished musculoskeletal function, individuals with CP suffer a high rate of moderate to severe bone fractures, which can lead to further immobility. Optimizing muscle and bone health with exercise may be important in minimizing fractures from limited mobility, and fundamental for maximizing health-related quality of life. The main purpose of this research is to investigate the effect of exercise training on musculoskeletal system in individuals with CP, with the goal of reducing the incidence of falls and fractures. To accomplish these aims, musculoskeletal health will be assessed using various physiological techniques (e.g., Dual energy X-ray Absorptiometry, Humac Norm Isokinematic System, Biodex Balance System) before, during, and after one year of exercise training in individuals with CP. In addition, various functional mobility tests to quantify fitness levels will be performed. Findings may lead to the development of novel therapeutic interventions targeted at improving musculoskeletal health in individuals with CP.

ELIGIBILITY:
Inclusion Criteria:

* those who can follow simple commands and walk independently with or without the use of an assistance apparatus (within Classification level I-III, based on Gross Motor Functioning Classification System, GMFCS) and have cerebral palsy will be included in the study. The rationale for such inclusion criteria (level I-III) is to make sure they can perform some leg exercise and tests.

Exclusion Criteria:

* If subjects have a history or symptoms of cardiovascular, renal, hepatic, or respiratory diseases, they will be excluded in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Height measurement | 1 minute
  Height (cm) will be measured using a standard beam scale with height rod. This anthropometric measurement is used to assess general body size. Body mass index is calculated and reported.
Body composition | 8 minutes
  Whole body Dual energy X-ray absorptiometry (DXA) will be measured to assess overall body composition for the mass of the bone, muscle, and fat in the whole body. For those who do not complete DXA due to severe spasticity, a bioelectrical impedance technique (BIA) using 4 electrode unit Biodynamics Model 310 Body Composition Analyzer will be used to quantify fat mass, fat free mass, and water content. BIA does not use x-ray; thus, participants will not be exposed additional radiation.
Muscular strength | 15 minutes
  Participants will perform leg press, leg curl, and leg extension at submaximal level to predict 1-Repetition Masimum using Brzycki equations. In addition, participants will perform knee extension and flexion testing using Humac Norm Isokinetic Dynamometer to measure isometric and isokinetic muscular strength in hamstrings and quadriceps.
Balance and related fall risks | 20 minutes
  Berg Balance Scale and Biodex Balance System will be used to assess balance and related fall risks. The Berg Balance Scale is a valid and reliable tool to assess populations with gait and balance issues. By completing 14 assessments with varying multiple tasks, participants will receive a point per task to have a final score which indicate the balance and risk of fall. Biodex Balance System assesses neuromuscular control by quantifying the ability to maintain dynamic bilateral and unilateral postural stability on both static and unstable surface. These tests will provide a quantified value for fall risk screening and conditioning status.
Bone mineral density | 8 minutes
  Bone mineral content and density using regional Dual energy X-ray absorptiometry (DXA) will be measured at regions of lumbar spine (L2-4), proximal femur at the hip joint, and forearm. T- and Z-scores of each region will be calculated to detect bone mineral density as well as the changes due to the intervention.
Weight measurement | 1 minute
  Weight (kg) will be measured using a standard beam scale with height rod. This anthropometric measurement is used to assess general body size. Body mass index is calculated and reported.
Waist and hip circumferences | 2 minutes
  Waist and hip circumference (cm) will be measured using a measuring tape. These anthropometric measurements are used to assess general body size.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abousalem, Ph.D, Study Director — SJSU
Locations (1):
- San Jose State University, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We understand the importance of data sharing and archiving for our scholarly community and to society at large. We are willing to share our data as for a significant contribution to the scientific community. Upon request, we will submit an share our data with public as recommended. However, as a part of informed consent process and to meet the confidentiality, we will not share any personal information of our research participants
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available 2 years after our manuscripts are published and for additional 3 years.
Access Criteria: Access to Individual Patient Data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan as well as the execution of a Data Sharing Agreement. For more information or to submit a request, please contact areum.jensen@sjsu.edu

DOCUMENTS (1):
  • Informed Consent Form (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT05070117/ICF_000.pdf